CLINICAL TRIAL: NCT00627848
Title: Effect of Rivastigmine on FMRI in Mild Alzheimer's Disease
Brief Title: Rivastigmine in Mild Alzheimer's Disease, FMRI Study
Acronym: ADFRMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Hilkka Soininen, Professor, Kuopio University Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: KUH5772749
Record Dates: First submitted 2008-02-22; First posted 2008-03-03 (Estimated); Last update posted 2011-10-28 (Estimated); Status verified 2011-10

CONDITIONS: Alzheimer' Disease
Keywords: Alzheimer's disease; fmri; face recognition; rivastigmine
MeSH Terms: conditions — Alzheimer Disease | interventions — Rivastigmine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: rivastigmine — Acute dose 3 mg or placebo. Thereafter 1.5 mg x 2 ad 30 days and thereafter increasing the dose upto 4.5 mg x 2 according to instructions.

SUMMARY:
The purpose of the study is to investigate the effect of rivastigmine given as an acute dose compared to placebo and after 1 month chronic dosing on fMRI response during a face recognition task. Furthermore, the aim is to investigate whether fMRI response is correlated with long term treatment effect at 6 months and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Probable Alzheimer's disease according to the NINCDS-ADRDA criteria
* mild disease, CDR 1
* the clinician is planning to start anticholinesterase treatment

Exclusion Criteria:

* cognitive impairment for other reason than Alzheimer's disease
* severe depression
* other unstable physical disease
* medal in body prevention MRI examination, claustrophobia
* cardiac pacemaker
* other significant neurologic or psychiatric disease
* contraindication for anticholinesterase treatment

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
FMRI response in face recognition task | at baseline and at 1 mo

SECONDARY OUTCOMES:
treatment response measured by ADAS-cog | at 6 month and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hilkka Soininen, Principal Investigator — Kuopio University Hospital
Locations (1):
- Kuopio University Hospital, Kuopio, Finland